CLINICAL TRIAL: NCT05845229
Title: Bioavailability of N-acylethanolamines: an Ileostomy Study.
Brief Title: Bioavailability of N-acylethanolamines: an Ileostomy Study (NAE Study)
Acronym: NAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REC/19/0096
Record Dates: First submitted 2023-02-28; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy Nutrition
Keywords: Lipid mediators; Nutrient sensing,; Bioavailability,; N-acylethanolamines,; Satiety.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-N-acylethanolamines meal (Experimental): Milk (150 mL), white bread (46 g), jam (10 g), cocoa powder (15 g), whole-grain cereals (30 g).
  Interventions: Dietary Supplement: High-N-acylethanolamine meal
- Low-N-acylethanolamines meal (Active Comparator): Milk (150 mL), whole-grain bread (80 g), jam (10 g), butter (5 g), instant coffee (2 g), dried apples (30 g).
  Interventions: Dietary Supplement: Low-N-acylethanolamine meal

INTERVENTIONS:
Dietary Supplement: High-N-acylethanolamine meal — Milk (150 mL), white bread (46 g), jam (10 g), cocoa powder (15 g), whole-grain cereals (30 g).
  Arms: High-N-acylethanolamines meal
Dietary Supplement: Low-N-acylethanolamine meal — Milk (150 mL), whole-grain bread (80 g), jam (10 g), butter (5 g), instant coffee (2 g), dried apples (30 g).
  Arms: Low-N-acylethanolamines meal

SUMMARY:
The endocannabinoids (ECs) and N-acylethanolamines (NAEs) are a group of endogenous lipid mediators which have a pleiotropic activity in the body modulating several biological pathways such as: appetite cues, food intake, blood pressure, inflammation, glycaemia, cognition and immunity. The ECs consist of N-arachidonoylethanolamide (AEA) and 2-arachidonoylglycerol (2-AG). They may have agonist activity on cannabinoid receptors CB1 and CB2 which are located in the central nervous system (CNS) and in peripheral tissues such as in the enteric nervous system (ENS), in the liver and in the adipose tissue. NAEs are known as "endocannabinoid-like" molecules and include oleoylethanolamine (OEA), linoleylethanolamine (LEA), and palmitoyletahanolamine (PEA). Evidence indicates that diet composition may affect fasting and post-prandial plasma ECs, N-acylphosphatidylethanolamines (NAPEs) and NAEs profile due to the content of their precursors, fatty acids and amines.

It is hypothesized that the concentration of NAPEs, NAEs and ECs in a meal could influence the intestinal concentrations of these lipid mediators that could bind the receptors located on the intestinal mucosa and in turn, differently modulate appetite and energy metabolism.

The study is an acute randomized crossover feeding study in ileostmists (n=14), having a breakfast meal low or high in NAPEs, NAEs and ECs. The meals are designed on a database published by our collaborators (University of Naples) and detailed in the research proposal. Concentrations of NAEs and ECs in urine, plasma and ileal fluid, beside the blood glucose, hormonal response, appetite feelings and food intake will be monitored over the experimental days.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have previously undergone an ileostomy and be more than 1.5-years post-operative
* Male or female
* Aged 18-70 years at recruitment

Exclusion Criteria:

* Participants not undergone an ileostomy and/or is less 1.5-years post-operative
* Adults <18 or >70 years at recruitment
* Pregnant/lactating female
* Current smokers
* Lactose intolerant
* Allergic to nuts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
N-acylphosphatidylethanolamines (NAPEs) levels in biofluids | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Significant changes from baseline in plasma, urines and, Ileal fluids levels of NAPEs by HPLC-MS analysis.
N-acylethanolamines (NAEs) levels in biofluids | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Significant changes from baseline in plasma, urines and, Ileal fluids levels of NAEs by HPLC-MS analysis.
Endocannabinoids levels in biofluids | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Significant changes from baseline in plasma, urines and, Ileal fluids levels of ECs by HPLC-MS analysis.

SECONDARY OUTCOMES:
Glycaemia | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of glycaemia by using a bedside glucometer.
Appetite sensations | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Significant changes from baseline in hunger, satiety, fullness and prospective of consumption.
Glucagon-like peptide 1 (GLP-1) plasmatic levels | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of GLP-1 by using of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Glucose-dependent insulinotropic peptide (GIP) plasmatic levels | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of GIP by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Insulin plasmatic levels | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of insulin by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Glucagon plasmatic levels. | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of glucagon by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
C-peptide plasmatic levels. | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of c-peptide by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Ghrelin plasmatic levels. | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of ghrelin by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Leptin plasmatic levels | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Measure of leptin by mean of Luminex kits in plasma samples pre-treated with protease inhibitor cocktail.
Energy intake during a buffet meal test | 0 hours
  Kilojoules
Gut microbiota composition | Change from baseline at 2, 4, 6 and, 8 hours after breakfast intake
  Microbiota composition will be determined by high throughput sequencing of the 16S ribosomal ribonucleic acid (rRNA) gene. The massive number of sequences obtained will be analyzed by using state of the art bioinformatics tools and the presence and relative abundance of the microbial species occurring in each sample will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No